CLINICAL TRIAL: NCT03990545
Title: Vessel Wall MR Imaging to Explore Sex-Differences of Intracranial Arterial Wall Changes After Suspected Stroke
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Jae W. Song, MD, MS, Jae W. Song, MD, Principal Investigator, University of Pennsylvania
Other Study IDs: 831803
Record Dates: First submitted 2019-06-14; First posted 2019-06-19 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Intracranial Atherosclerosis; Acute Stroke; Transient Ischemic Attack
Keywords: intracranial atherosclerotic disease; acute stroke; transient ischemic attack; vessel wall imaging
MeSH Terms: conditions — Intracranial Arteriosclerosis; Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cases with stroke
- Controls without stroke

SUMMARY:
Despite advances in stroke care, women continue to face worse outcomes after stroke than men. This disparity in outcomes may be related to biologic sex-differences that manifest in the development and progression of atherosclerosis. Decades of cyclic changes in the hormonal milieu lead to different metabolic profiles in women. These changes may also explain sex-differences in risk factor profiles of atherogenesis and plaque composition. The investigators' objective is to conduct a cross-sectional MR imaging study of suspected stroke patients to compare the burden and composition of intracranial atherosclerosis and risk factors between men and women. Results from this study are expected to show that sex and sex-specific risk factors should be considered at the outset of stroke evaluation for risk-stratification. In the era of precision medicine, the investigators propose the role of sex should be a starting point in the clinical evaluation of stroke.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Suspected stroke patients
* No contraindications for an MRI exam or gadolinium intravenous contrast
* No need for an emergent interventional treatment (e.g., thrombectomy)

Exclusion Criteria:

* Younger than 18 years
* Pregnant

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Suspected stroke patients
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2021-03-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of intracranial arterial wall abnormalities by sex. | 1 day (Evaluated at time of clinical presentation).
  Vessel wall imaging characteristics on multicontrast MR imaging

CONTACTS AND LOCATIONS:
Overall Officials: Jae W Song, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States